CLINICAL TRIAL: NCT07142655
Title: Post-Marketing Database Study for Rivaroxaban in Patients With PAD After Lower Limb Revascularization.
Brief Title: An Observational Study to Learn More About the Safety of Rivaroxaban in Participants With Peripheral Arterial Disease Who Had Surgery to Improve Blood Flow to Their Legs
Status: Active, not recruiting | Type: Observational
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Other Study IDs: 22340
Record Dates: First submitted 2025-08-25; First posted 2025-08-27 (Actual); Last update posted 2025-10-08 (Actual); Status verified 2025-10

CONDITIONS: Peripheral Arterial Disease (PAD)
MeSH Terms: conditions — Peripheral Arterial Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Exposure: Patients who were prescribed rivaroxaban 2.5 mg during the enrollment period
- Reference: Patients who were not prescribed rivaroxaban 2.5mg during the enrollment period and were matched with patients in the exposure group

SUMMARY:
This is an observational study in which data already collected from people with peripheral arterial diseases (PAD) who had a surgery to improve blood flow to their legs are studied.

The study is conducted to check the safety of rivaroxaban after it is approved and available in Japan.

In observational studies, only observations are made without participants receiving any advice or changes to healthcare.

PAD is a condition where blood flow is reduced in the arteries of the legs and arms. This can cause pain, numbness, or weakness in the legs, and increases the risk of heart attack and other heart-related problems. People with PAD may undergo surgery to improve blood flow to their legs, in which doctors use a thin tube to open a narrow or blocked blood vessel in the legs.

The study drug, rivaroxaban, is already approved for doctors to prescribe to people with PAD. It works by blocking a protein that causes blood clots, helping to prevent clot formation and improving blood flow.

The participants in this study are already receiving treatment with rivaroxaban 2.5 milligrams (mg) as part of their regular care from their doctors.

There have been studies in which researchers studied the effect and safety of rivaroxaban in participants with PAD who had a surgery to improve blood flow to their legs. However, these studies included only a small number of Japanese participants. In this study, researchers will specifically gather data from Japanese participants to further understand the safety of rivaroxaban.

The main purpose of the study is to learn more about the safety of rivaroxaban 2.5 mg in Japanese participants with PAD who had a surgery to improve blood flow to their legs.

To do this, researchers will collect information about:

* any bleeding event participants have had during their treatment with rivaroxaban
* the participants who died due to the heart and blood flow related problems while receiving rivaroxaban, compared to those who did not receive it

The data will come from electronic healthcare records for people in Japan who had a surgery to improve blood flow to their legs and were diagnosed with PAD between October 2021 to September 2025.

In this study, only available data from routine care are collected. No visits or tests are required as part of this study.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with PAD in or before the month following the index date
* Lower limb revascularization was performed in or before the month of PAD diagnosis
* Age 18 years or older as of the index date

Exclusion Criteria:

* Lower limb revascularization performed in the same month or before the month of PAD diagnosis was performed after the index date
* Index date before the start date of the enrollment period

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population is patients with PAD after lower limb revascularization.
Sampling Method: Probability Sample
Enrollment: 1500 (Actual)
Dates: Start 2025-08-12 (Actual); Primary Completion 2025-10-31 (Estimated); Study Completion 2025-10-31 (Estimated)

PRIMARY OUTCOMES:
Hemorrhage requiring for blood transfusion | Retrospective analysis from 01-OCT-2021 to 30-SEPT-2025
  If all of the following criteria are met:
  * A transfusion with a blood volume equivalent to > 800 mL is recorded after the index date
  * No surgery other than endoscopic hemostasis surgery is performed on the day before or on the day of the transfusion
  * No anticoagulants is prescribed on the day following the transfusion
Intracranial bleeding | Retrospective analysis from 01-OCT-2021 to 30-SEPT-2025
  If all of the following criteria are met:
  * An Magnetic Resonance Imaging (MRI) or a Computed Tomography (CT) examination is performed at or after the index date
  * A diagnosis for any intracranial bleeding is recorded in the same month of the MRI or CT examination
  * A rehabilitation for stroke or a death is recorded within 30 days after the MRI or CT examination
Intraocular bleeding | Retrospective analysis from 01-OCT-2021 to 30-SEPT-2025
  If all of the following criteria are met:
  * An ophthalmologic examination is performed after the index date
  * A diagnosis for any intraocular bleeding is recorded in the same month of the ophtalmologic examination
Upper gastrointestinal bleeding | Retrospective analysis from 01-OCT-2021 to 30-SEPT-2025
  If all of the following criteria are met:
  * An examination related to an upper gastrointestinal bleeding is performed after the index date
  * A diagnosis for any upper gastrointestinal bleeding is recorded in the same month of examination
  * No anticoagulants is prescribed on the day following the examination
Lower gastrointestinal bleeding | Retrospective analysis from 01-OCT-2021 to 30-SEPT-2025
  If all of the following criteria are met:
  * An examination related to a lower gastrointestinal bleeding is performed after the index date
  * A diagnosis for any lower gastrointestinal bleeding is recorded in the same month of examination
  * No anticoagulants is prescribed on the day following the examination
Sudden cardiac death | Retrospective analysis from 01-OCT-2021 to 30-SEPT-2025
  A diagnosis for sudden cardiac death is recorded after the index date.
Acute coronary syndrome and death | Retrospective analysis from 01-OCT-2021 to 30-SEPT-2025
  If all of the following criteria are met:
  * A diagnosis for Acute coronary syndrome is recorded after the index date
  * At the date of sudden cardiac death, Peripheral Component Interconnect (PCI) is recorded
  * Death within 30 days of sudden cardiac death

SECONDARY OUTCOMES:
All cause death | Retrospective analysis from 01-OCT-2021 to 30-SEPT-2025
  Date of death. A diagnosis for death related disease or death is recorded after the index date. The index date is defined as:
  * The date of the first prescription of rivaroxaban 2.5mg during the enrollment period (from 24-OCT-2022 to 30-SEP-2025), for patients included in the exposure group.
  * The earliest date of prescription of either aspirin or clopidogrel after the date of lower limb revascularization, for patients included in the reference group
Re-performing lower limb revascularization | Retrospective analysis from 01-OCT-2021 to 30-SEP-2025
  Date of lower limb revascularization. In case of multiple lower limb revascularizations, the earliest date after the index date will be used. The index date is defined as:
  * The date of the first prescription of rivaroxaban 2.5mg during the enrollment period (from 24-OCT-2022 to 30-SEP-2025), for patients included in the exposure group.
  * The earliest date of prescription of either aspirin or clopidogrel after the date of lower limb revascularization, for patients included in the reference group

CONTACTS AND LOCATIONS:
Locations (1):
- Medical Data Vision Co., Ltd, Tokyo, Japan

IPD SHARING:
Plan to Share IPD: No
Availability of this study's data will later be determined according to Bayer's commitment to the EFPIA/PhRMA "Principles for responsible clinical trial data sharing". This pertains to scope, timepoint and process of data access. As such, Bayer commits to sharing upon request from qualified researchers patient-level clinical trial data, study-level clinical trial data, and protocols from clinical trials in patients for medicines and indications approved in the US and EU as necessary for conducting legitimate research. This applies to data on new medicines and indications that have been approved by the EU and US regulatory agencies on or after January 01, 2014. Interested researchers can use www.vivli.org to request access to anonymized patient-level data and supporting documents from clinical studies to conduct research. Information on the Bayer criteria for listing studies and other relevant information is provided in the member section of the portal.